CLINICAL TRIAL: NCT06025786
Title: Impact Assessment of Benazir Nashonuma Program (BNP) on Stunting Prevention Among Children 0-59 Months of Age in Pakistan
Brief Title: Impact Evaluation of Benazir Nashonuma Program (BNP) on Stunting Among Under-five Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: International Food Policy Research Institute (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Distinguished University Professor and Founding Director of the Institute for Global Health and Development and the Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BNP Quasi Experimental Study
Record Dates: First submitted 2023-08-16; First posted 2023-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-07

CONDITIONS: Stunting; Wasting; Anemia; Nutrient Deficiency
Keywords: Quasi experimental study; Maternal and child nutrition; Stunting; Wasting; Under-five malnutrition; Specialized Nutritious Food (SNF)
MeSH Terms: conditions — Growth Disorders; Cachexia; Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Districts with established and operational BNP implementation (Experimental): The intervention arm consists of nine districts from four provinces and two regions of Pakistan where the Benazir Nashonuma Program (BNP) is operational, providing reproductive and healthcare services to pregnant women and their children under the age of two.
  Interventions: Combination Product: Benazir Nashonuma Program (BNP)
- Districts without BNP implementation and functionality (No Intervention): The control arm comprises of nine districts where Benazir Nashonuma Program (BNP) has not been implemented. These districts are comparable to their respective intervention districts in terms of average maternal BMI and prevalence of stunting.

INTERVENTIONS:
Combination Product: Benazir Nashonuma Program (BNP) — Benazir Nashonuma Program (BNP)
  Dietary supplement for pregnant women and lactating mothers during the first six months of lactation:
  Maamta is a 75-gram sachet made from peanut butter with 400 kcal of energy
  Dietary supplement for children aged 6-23 months:
  Wawamum is a lipid-based nutrient supplement consisting of skimmed milk powder, micronutrients, vegetable oil, roasted chickpeas and antioxidants. Wawamum covers the recommended daily dose of most micronutrients and 255 kcal of energy.
  Conditional Cash Transfer (CCT):
  This includes stipends of PKR 2000 during pregnancy contingent on three antenatal care visits, consuming SNF, attending awareness sessions on health and nutrition, getting two doses of tetanus toxoid and institutional delivery. After delivery PKR 2000/- for boys and 2500/- for girls are paid as incentives conditioned on getting child's birth registered, routine immunization and consumption of SNF by the child from 6-23 months
  Arms: Districts with established and operational BNP implementation

SUMMARY:
The aim of the study is to evaluate the impact of Benazir Nashonuma Program (BNP) on prevalence of stunting among under-five children in low income setting of Pakistan. The research question that the study aims to answer is:

Is there any change in the prevalence of stunting among under-five children in districts where Benazir Nashonuma Program (BNP) is established compared to districts where BNP is not established?

Districts where BNP is functional, and women and children are receiving the intervention will be compared at baseline and end line with control districts where conventional reproductive care services are given. Prevalence of stunting among under-five children will be compared along with other nutritional and growth status indicators over a period of 4 years.

DETAILED DESCRIPTION:
Maternal and child malnutrition is a significant public health challenge, with 40% of under five children being stunted in Pakistan. Stunting is associated with morbidity and mortality with detrimental effects on the physical, social and cognitive development of children. The two key determinants include maternal undernutrition during in-utero and poor infant and child feeding practices in the first two years of life. The opportunity to improve maternal, infant, and child outcomes is provided by the interventions aimed at improving maternal and child nutrition throughout the first 1000 days, known as "window of opportunity". In this study, the investigators aim to assess the effectiveness of the Benazir Nashonuma Programme (BNP) on stunting reduction and related maternal and child health outcomes and to determine the uptake of BNP related services in the intervention districts in all provinces and regions of Pakistan.

The study will achieve the following objectives:

Primary Objective

• To determine the baseline to end-line change in the prevalence of stunting among children 0-59 months of age among low income settings

Secondary Objectives

For under-five children:

To determine the baseline to end-line change in the

* Prevalence of wasting among children 0-59 months of age
* Prevalence of underweight children 0-59 months of age
* Prevalence of Moderate Acute Malnutrition (MAM) among children 0-59 months of age
* Prevalence of Severe Acute Malnutrition (SAM) among children 0-59 months of age
* Prevalence of 0-23 months old children meeting Infant and Young Child Feeding (IYCF) indicators including exclusive breastfeeding, complementary feeding, dietary diversity, minimum acceptable diet and minimum meal frequency.
* Proportion of children 0-59 months of age who received all recommended vaccinations according to the national immunization schedule.

For Women of Reproductive Age (15- 49 years):

To determine the baseline to end-line change in the

* BMI (body mass index) and prevalence of underweight women of reproductive age (WRA)
* Reproductive services uptake by WRA
* Minimum dietary diversity among WRA
* Percentage of households that experienced food insecurity.

A quasi-experimental study with baseline and end-line cross-sectional surveys will be conducted in 18 districts of the four provinces and two administrative areas of Pakistan. The intervention districts includes Shaheed Benazir Abad and Dadu from Sindh, Rajanpur from Punjab, Lasbela and Harnai from Balochistan, Upper Dir and Tank from Khyber Pakhtunkhwa, Diamer from Gilgit Baltistan and Bagh from Azad Jammu and Kashmir. Their control districts are Sangarh, Naushero Feroze, Bahawalnagar, Sibbi, Sherani, Shangla, D. I. Khan, Shigar and Muzaffarbad respectively.

The study will employ a two-stage cluster sampling to enroll children 0-59 months of age and their mothers/caregivers from the 13,200 households (734 per district). The primary (PSUs) and secondary sampling units (SSUs) will include villages and households respectively.

ELIGIBILITY:
All those households are eligible to be included in the study who have:

* An under-five child with a mother registered with Benazir Income Support Program (BISP)
* Both available at the time of interview

Exclusion criteria includes:

• Mother of the child who is not a woman of reproductive age, i.e., less than 15 years or greater than 49 years

Ages: 1 Day to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline to end-line change in the prevalence of stunting among children 0-59 months of age | 3 years (on study completion)
  Height-for-age ≤-2 SD of the WHO Child growth standards median

SECONDARY OUTCOMES:
Baseline to end-line change in the prevalence of underweight women of reproductive age (15-49 years) | 3 years (on study completion)
  WRA with a Body Mass Index (BMI) less than 18.5 kg/m2 will be considered underweight
Baseline to end-line change in the prevalence of wasting among children 0-59 months of age | 3 years (on study completion)
  Weight-for-height ≤-2 SD of the WHO Child growth standards median
Baseline to end-line change in the prevalence of food insecurity status at household level | 3 years (on study completion)
  Food Insecurity Experience Scale (FIES) by Food and Agriculture Organization (FAO) is experience-based measures of household or individual food security. It consists of eight questions regarding people's access to adequate food in last 12 months due to lack of money or other resources. Food insecurity is reported as mild, moderate and severe.
Baseline to end-line change in the number of antenatal care (ANC) visits during pregnancy | 3 years (on study completion)
  Number of antenatal care (ANC) visits done during the preceding pregnancy, leading to a live birth within the last two years.
Baseline to end-line change in the prevalence of institutional deliveries | 3 years (on study completion)
  Number of women who gave birth at a healthcare facility during the preceding pregnancy, leading to a live birth within the last two years.
Baseline to end-line change in the prevalence of skilled birth attendance | 3 years (on study completion)
  Number of women whose birth was attended by a skilled health personnel during the preceding pregnancy, leading to a live birth within the last two years.
Baseline to end-line change in prevalence of utilization of iron folic acid (IFA) during pregnancy | 3 years (on study completion)
  Consumption of iron folic acid tablets during pregnancy
Baseline to end-line change in the prevalence of Minimum dietary diversity for women (MDDW) | 3 years (on study completion)
  Consumption of at least five out of the ten food groups during the previous day and night (24 hours)
Baseline to end-line change in the prevalence of infants who were ever breastfed | 3 years (on study completion)
  Number of infants who were breastfed at least once
Baseline to end-line change in the prevalence of exclusive breastfeeding among infants 0-5 months of age | 3 years (on study completion)
  Number of infants who were fed exclusively with breast milk during the previous day

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, PhD, FRC, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Muhammad S, Malik AA, Soofi S, Habib A, Umer M, Rizvi A, Ahmed I, Leroy J, Cousens S, Bhutta ZA. Impact assessment of Benazir Nashonuma Programme (BNP) on maternal, child health and nutritional status in Pakistan: a quasi-experimental study protocol. BMJ Open. 2025 Jun 27;15(6):e094565. doi: 10.1136/bmjopen-2024-094565. PMID 40578861